CLINICAL TRIAL: NCT01944852
Title: Efficacy and Safety of a Double Icodextrin Dose in Elderly Incident CAPD Patients on Incremental Peritoneal Dialysis Therapy: the DIDo Study
Brief Title: Efficacy and Safety of a Double Icodextrin Dose in Elderly Incident CAPD Patients on Incremental PD.
Acronym: DIDo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pr Eric Goffin (Other)
Responsible Party: Sponsor-Investigator, Pr Eric Goffin, Professor, Université Catholique de Louvain
Organization: Université Catholique de Louvain (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL_2011_DIDo
Record Dates: First submitted 2013-09-02; First posted 2013-09-18 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Renal Insufficiency
Keywords: icodextrin; double dose; elderly incident CAPD patients; DIDo study
MeSH Terms: conditions — Renal Insufficiency | interventions — Icodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 icodextrin bags/day (Experimental): 2 icodextrin bags + 1 glucose per day
  Interventions: Drug: Icodextrin
- 1 icodextrin bag/day (Active Comparator): 1 icodextrin bag + 2 glucose bags per day
  Interventions: Drug: Icodextrin

INTERVENTIONS:
Drug: Icodextrin
  Other Names: Extraneal

SUMMARY:
The DIDo study is an open-label, randomised, multicentre study with 2 parallel groups in incident CAPD patients aged of 65 at minimum :

* One group in which patients will receive 2 bags of icodextrin/day and 1 bag of glucose
* One group in which patients will receive 1 bag of icodextrin/day and 2 bags of glucose.

DETAILED DESCRIPTION:
The DiDo study evaluates efficacy and safety of a Double Icodextrin Dose in elderly incident CAPD patients on incremental Peritoneal Dialysis therapy.

The objective is to demonstrate the superiority and safety of using 2, as compared to 1, icodextrin bags / day, in a cohort of elderly incident continuous ambulatory peritoneal dialysis (CAPD) patients using incremental peritoneal dialysis (PD) (3 bags / day), with the aim of prolonging the period of time for which incremental PD can be used.

This is a phase IV open-label, randomised, multicentre study with 2 parallel groups, which will take place in up to 30 hospital out-patient clinics un Europe.

It is planned to include 160 patients on the run-in period in order to obtain 100 randomised patients and 90 patients evaluable at the primary endpoint (45 in each group). The duration of patient recruitment is estimated at 1 year but this may be extended until all 160 patients are recruited.

There are 2 periods: a run-in period of 2 months and a treatment period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

Run-in period

* Incident CAPD patients who require incremental PD and in whom a 1.5L dialysate can be safely instilled,
* Creatinine clearance < 20 ml / min (calculated with the modification of the Diet in renal Disease [MDRD] formula),
* Age ≥ 60 years,
* Patients willing and able to give written informed consent and comply with the requirements of the study protocol.

Treatment period

* Patients having successfully completed the run-in period (achieving euvolemia)

Exclusion Criteria:

Run-in period

* Contraindication for CAPD according to local practice,
* Life expectancy < 6 months,
* Known allergy to icodextrin (cloudy dialysate or skin rash),
* Need for amino-acid prescription,
* Treatment with any investigational product within 30 days prior to signature of the informed consent form (ICF)
* History of drug or alcohol abuse within 3 months prior to the signature of the ICF.

Treatment period

* Severe symptomatic arterial hypotension at the end the run-in period in the Investigator's opinion,
* Excessive ultrafiltration (UF) during the run-in period,
* Allergy to icodextrin discovered during the run-in period,
* Impossibility to achieve adequate PD regimen within the run-in period (catheter dysfunction, peritoneal leaks, inadequate compliance, psychosocial reasons)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients stopping 3 bags / day | During the treatment phase of 18 months
  The primary endpoint will be the proportion of patients stopping 3 bags / day for the following reasons:
  * Use of > 15 % hypertonic glucose dialysate 3.86 % or > 30 % hypertonic glucose dialysate 2.27 % over a 4-week period19-20,
  * Transfer of the patient to another dialysis method (HD, APD, CAPD with > 3 bags / day) for any reason,
  * Death of the patient.

SECONDARY OUTCOMES:
effect on clinical and biological determinants | During 18 months, evaluated on month 3, 6, 9, 12 and 18.
  • Metabolic control: HbA1c and lipid concentration (total, high-density lipoprotein [HDL], low-density lipoprotein [LDL], triglycerides, cholesterol)
effect on clinical and biological determinants | During 18 months, evaluated on month 3, 6, 9, 12 and 18.
  • Blood pressure control, evaluated by the number of anti-hypertensive agents and daily furosemide dose, and measured at the end of each study visit
effect on clinical and biological determinants | During 18 months, evaluated on month 3, 6, 9, 12 and 18.
  • Nutritional aspect: serum albumin and prealbumin concentrations based on the changes in percentage at various time points compared to baseline (V2)
effect on clinical and biological determinants | During 18 months, evaluated on month 3, 6, 9, 12 and 18.
  • Inflammatory profile: CRP concentrations
effect on clinical and biological determinants | Month 9 and month 18.
  • Left ventricular mass calculated following echocardiography
effect on clinical and biological determinants | Month 6, 12 and 18.
  • Quality of life according to KDQoL
effect on clinical and biological determinants | During 18 months, evaluated on month 3, 6, 9, 12 and 18.
  • Residual renal function evaluated by calculated GFR
effect on clinical and biological determinants | On month 6, 12 and 18.
  • Peritoneal membrane permeability assessed by the PET
effect on clinical and biological determinants | During the treatment phase of 18 months.
  • Number of hospitalisations and length (in days) of hospitalisation
Safety endpoints | Durign the treatment phase of 18 months.
  • Adverse events (AEs), treatment-emergent AEs and serious adverse events (SAEs)
6.1.3 Safety endpoints | On month 3, 6, 12 and 18.
  • Serum sodium concentration and icodextrin metabolites concentration
safety endpoints | During the treatment phase of 18 months.
  • Relevant clinical problems related to serum sodium concentration and to icodextrin metabolites accumulation
Safety endpoints | During the treatment phase of 18 months.
  • Incidence of skin rashes
Safety endpoints | During the treatment phase of 18 months.
  • Incidence of sterile peritonitis

CONTACTS AND LOCATIONS:
Overall Officials: Eric Goffin, Principal Investigator — UCL
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Morelle J, Lambie M, Oberg CM, Davies S. The Peritoneal Membrane and Its Role in Peritoneal Dialysis. Clin J Am Soc Nephrol. 2024 Feb 1;19(2):244-253. doi: 10.2215/CJN.0000000000000282. Epub 2023 Aug 24. PMID 37616463